CLINICAL TRIAL: NCT02056652
Title: Prevention of Preterm Birth With a Pessary in Singleton Gestations
Acronym: PoPPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 817797
Record Dates: First submitted 2014-02-04; First posted 2014-02-06 (Estimated); Results first posted 2018-05-29 (Actual); Last update posted 2018-05-29 (Actual); Status verified 2018-04

CONDITIONS: Preterm Birth; Short Cervix
Keywords: Preterm birth; Preterm delivery; short cervix; pessary
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pessary (Experimental): Use of the Bioteque cup pessary. Pessary will be placed between 18 and 23 6/7 weeks gestation, and will be removed during the 37th week of pregnancy (or earlier, if indicated)
  Interventions: Device: Bioteque cup pessary
- No pessary (No Intervention): No pessary will be used. Subjects will receive standard obstetrical management

INTERVENTIONS:
Device: Bioteque cup pessary
  Arms: Pessary

SUMMARY:
Preterm birth (PTB) is associated with over one million infant deaths annually worldwide. The incidence of PTB in the United States is 11.5% with more than 500,000 deliveries occurring at less than 37 weeks gestation annually. The rate of PTB in the United States increased to 12.8% in 2006, and remains high compared to almost all other developed countries, despite the introduction of many public health and medical interventions designed to delay PTB. Weekly treatment with 17-alpha hydroxyprogesterone caproate beginning at 16-20 weeks gestation has been shown to significantly reduce the risk of PTB and is currently recommended for women who experienced spontaneous PTB in a prior pregnancy. However, a strategy for the prevention of spontaneous PTBs in which therapeutic intervention is restricted to women with a previous PTB is likely to have a small effect on the overall rate of prematurity since only about 10% of spontaneous PTBs arise in women with such a history. A major reduction in rates of mortality and morbidity in premature babies will only be achieved with increased precision in the identification of women at risk of spontaneous PTB and through the development of an effective prevention for this complication. Transvaginal ultrasound measurement of cervical length is a reliable screening test for prediction of PTB. Although treatment with vaginal progesterone is effective in decreasing PTB in women with a short cervix, over 30% of women still experience premature delivery and many women find daily administration of progesterone to be challenging. Preliminary studies have suggested that use of an intravaginal pessary may be effective in preventing PTB. If effective this approach would be particularly appealing because of the wide availability of pessaries, ease of use, and low cost. Unfortunately, existing studies are inadequate to confirm effectiveness; a well designed, properly powered, prospective randomized trial is warranted prior to widespread implementation in clinical practice. We propose such a trial to study the effectiveness of the pessary in decreasing the incidence of PTB in an inner city Philadelphia population.

ELIGIBILITY:
Inclusion Criteria:

* 18-50 years of age
* Singleton pregnancy (limits the participants to female gender)
* Short cervical length (less than or equal to 25 mm) on second trimester ultrasound at 18-23 6/7 weeks gestation

Exclusion Criteria:

* Multiple gestation
* Prior spontaneous preterm birth 16-36 6/7 weeks
* Ruptured membranes
* Lethal fetal structural anomaly
* Fetal chromosomal abnormality
* Cerclage in place (or planned placement)
* Vaginal bleeding
* Suspicion of chorioamnionitis
* Ballooning of membranes outside the cervix into the vagina or CL = 0 mm on transvaginal ultrasound
* Painful regular uterine contractions
* Placenta previa

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 122 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lorraine Dugoff, MD, Principal Investigator — University of Pennsylvania; Vincenzo Berghella, MD, Principal Investigator — Thomas Jefferson University; Jack Ludmir, MD, Principal Investigator — University of Pennsylvania
Locations (4):
- United States (4):
  - Geisinger Medical Center, Danville, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Abdel-Aleem H, Shaaban OM, Abdel-Aleem MA, Aboelfadle Mohamed A. Cervical pessary for preventing preterm birth in singleton pregnancies. Cochrane Database Syst Rev. 2022 Dec 1;12(12):CD014508. doi: 10.1002/14651858.CD014508. PMID 36453699

RESULTS

PARTICIPANT FLOW:
Groups:
- Pessary: Use of the Bioteque cup pessary. Pessary will be placed between 18 and 23 6/7 weeks gestation, and will be removed during the 37th week of pregnancy (or earlier, if indicated)
  Bioteque cup pessary
Period: Overall Study
Arm/Group | Pessary | No Pessary
Started | 61 | 61
Completed | 60 | 58
Not Completed | 1 | 3
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pessary | No Pessary | Total
Number analyzed (Participants) | 61 | 61 | 122
Age, Customized [Mean (Full Range); unit: years]
  Maternal Age | 27.7 [23.0 to 32.3] | 29.5 [23.0 to 34.8] | 28.6 [23.0 to 34.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 61 | 122
  Male | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 61 | 61 | 122

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Experiencing Preterm Birth
Description: Birth before 37 weeks gestation was captured.
Time Frame: Before 37 weeks gestation (20 0/7 - 36 6/7 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Pessary | No Pessary
Number analyzed (Participants) | 60 | 58
Participants | 26 | 23

2. Secondary Outcome: Average Birth Weight of Babies Born on Trial
Description: The birth weights of babies born in the pessary group was compared to those born in the no pessary group
Time Frame: Time of delivery
Measure: Mean (Full Range); unit: grams
Arm/Group | Pessary | No Pessary
Number analyzed (Participants) | 60 | 58
grams | 2788 [1285 to 3188] | 2843 [1035 to 3329]

3. Secondary Outcome: Number of Participants That Experienced Spontaneous Preterm Births on Trial
Description: The number of spontaneous births that occurred in participants on trial before 37 weeks was captured.
Time Frame: Before 37 weeks gestation
Measure: Count of Participants; unit: Participants
Arm/Group | Pessary | No Pessary
Number analyzed (Participants) | 60 | 58
Participants | 23 | 19

4. Secondary Outcome: Number of Participants Experiencing Spontaneous Rupture of Membranes
Description: Rupture of membranes before 34 weeks gestation was captured in each group.
Time Frame: Less than 34 weeks gestation
Measure: Count of Participants; unit: Participants
Arm/Group | Pessary | No Pessary
Number analyzed (Participants) | 60 | 58
Participants | 18 | 10

5. Secondary Outcome: Number of Subjects Experiencing Neonatal Death
Description: Number of participants who experienced neonatal deaths from birth to day 28 was captured for each group.
Time Frame: Between birth and 28 days of age
Measure: Count of Participants; unit: Participants
Arm/Group | Pessary | No Pessary
Number analyzed (Participants) | 60 | 58
Participants | 3 | 6

6. Secondary Outcome: Number of Subjects Experiencing Chorioamnionitis
Description: The AE of Chorioamnionitis was captured for each group.
Time Frame: Time of delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Pessary | No Pessary
Number analyzed (Participants) | 60 | 58
Participants | 7 | 4

ADVERSE EVENTS:
Arm/Group | Pessary | No Pessary
All-Cause Mortality (participants affected / at risk) | 0/61 | 0/61
Serious Adverse Events (participants affected / at risk) | 0/61 | 0/61
Other Adverse Events (participants affected / at risk) | 3/61 | 6/61
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pessary (N=61) | No Pessary (N=61)
Bacterial Vaginosis (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 6 (6) — BV was accessed in both groups

LIMITATIONS AND CAVEATS:
Our main limitation was the small sample size due to the fact that the study was stopped before planned enrollment was completed. In order to reach significance, we would need for the next 60 subjects randomized to the pessary group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No